CLINICAL TRIAL: NCT06359249
Title: Do the Symptoms of Chronic Constipation Improve With a Primary Care Programme Based on Behavioural Re-education and Abdominal Massage? A Randomised Control Trial
Brief Title: Do the Symptoms of Chronic Constipation Improve With a Primary Care Programme Based on Behavioural Re-education and Abdominal Massage?
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Universitat de Vic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V.3-06/02/2024
Record Dates: First submitted 2024-03-18; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Constipation Chronic Idiopathic
Keywords: Chronic constipation; abdominal massage; proctologic disease; pelvic floor disorders; physical therapy
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Habitual treatment
- behavioural intervention group (Experimental): Conductual treatment
  Interventions: Behavioral: change of habits
- behavioural intervention and massage group (Experimental): Conductual and abdominal massage treatment
  Interventions: Other: change of habits + auto abdominal massage

INTERVENTIONS:
Behavioral: change of habits — change of habits
  Arms: behavioural intervention group
Other: change of habits + auto abdominal massage — change of habits + auto abdominal massage
  Arms: behavioural intervention and massage group

SUMMARY:
Constipation is one of the most common digestive problems in today's society. In Spain, it is estimated that this condition affects between 12% and 20% of the population, being more frequent in women, contributing considerably to the quality of life, to the increase of medical visits and to high costs for the health system. The objectives of the study are to reduce the rate of constipation and laxative use in the short term with a structured rehabilitation programme consisting of abdominal massage therapy and behavioural re-education, to improve the quality of life of these patients, and to assess whether the proposed treatment is effective in the short and medium term.

DETAILED DESCRIPTION:
Background: Constipation is one of the most common digestive problems in today's society. In Spain, it is estimated that this condition affects between 12% and 20% of the population, being more frequent in women, contributing considerably to the quality of life, to the increase of medical visits and to high costs for the health system. The objectives of the study are to reduce the rate of constipation and laxative use in the short term with a structured rehabilitation programme consisting of abdominal massage therapy and behavioural re-education, to improve the quality of life of these patients, and to assess whether the proposed treatment is effective in the short and medium term.

Method: Randomised clinical trial. Participants: people with constipation in the region of L'Anoia, Catalonia. There will be 3 groups: the control group (CG), behavioural intervention group (BIG) and behavioural intervention and massage group (BIMG). Constipation will be assessed with the Bristol scale, Rome IV Criteria and the number of laxatives; and quality of life with the CVE-20 Questionnaire.

Participants will be proposed from Primary Care Centres in the region of L'Anoia, Catalonia, Spain.

Inclusion criteria:

* Having been diagnosed with primary constipation using Rome IV Criteria(11), of more than three months' duration.
* Understanding Catalan, Spanish or English.

Exclusion criteria:

* Having constipation secondary to neurogenic, metabolic, endocrine or postoperative diseases.
* Having constipation secondary to medication for other pathologies, the medication list for which can be found in the annex.
* Having any type of open abdominal and/or anal wound, such as a recent abdominal scar or anal fissure.
* Meeting any absolute contraindication criteria for the use of abdominal massage therapy, such as an unstable fracture requiring absolute rest and immobilisation, pregnancy or active oncological procedures.
* Suffering from some type of cognitive, psychiatric or neurological alteration that does not allow to understand the project.

Discussion: Research is needed on conservative, non-pharmacological treatment to try to reduce one of the main conditions affecting public health, and thus reduce the possible illnesses associated with constipation and reduce costs to the health system.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with primary constipation using Rome IV Criteria(11), of more than three months' duration.
* Understanding Catalan, Spanish or English.

Exclusion Criteria:

* Having constipation secondary to neurogenic, metabolic, endocrine or postoperative diseases.

  * Having constipation secondary to medication for other pathologies, the medication list for which can be found in the annex.
  * Having any type of open abdominal and/or anal wound, such as a recent abdominal scar or anal fissure.
  * Meeting any absolute contraindication criteria for the use of abdominal massage therapy, such as an unstable fracture requiring absolute rest and immobilisation, pregnancy or active oncological procedures.
  * Suffering from some type of cognitive, psychiatric or neurological alteration that does not allow to understand the project.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Degree of constipation | Day 0, Month 3, Month 6
  Degree of constipation with Rome IV Criteria
Stool characteristics | Day 0, Month 3, Month 6
  Stool characteristics with the Bristol Scale
Quality of life focused on patients with constipation | Day 0, Month 3, Month 6
  Quality of life focused on patients with constipation with the CVE-20 questionnaire from an emotional, physical and social viewpoint.
The number of laxatives taken by each participant | Month 3, Month 6
  The number of laxatives taken by each participant with an accounting schedule.

SECONDARY OUTCOMES:
Other patient characteristics such as sex, age, previous conditions, and level of physical activity with the VREM questionnaire. | Day 0, Month 3, Month 6

CONTACTS AND LOCATIONS:
Locations (1):
- Cristina Segura Bayona, Igualada, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No